CLINICAL TRIAL: NCT04128865
Title: PRevention of INteractions Between Phytotherapies and CancEr Treatments by a SmartphonE/Tablet Automated SurvEy
Acronym: PRINCESSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Paul Gougis (Other)
Responsible Party: Sponsor-Investigator, Paul Gougis, MD, Groupe Hospitalier Pitie-Salpetriere
Organization: Groupe Hospitalier Pitie-Salpetriere (Other)
Other Study IDs: CIC1421-18-07
Record Dates: First submitted 2018-04-10; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Cancer
Keywords: phytotherapy; dietary supplement; food interaction; herb-drug interactions
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The use of phytotherapies or specific food or dietary supplement (HFDS) is common among cancer patients. They can also be responsible of clinically relevant interaction with anti-cancer treatments. This study aims at assessing the proportion patients using HFDS which are likely to have an interaction with their anticancer treatments. The data is collected through a smartphone/tablet application. The aim of the study is to demonstrate that clinically significant herb-drug interaction with anticancer treatment could be avoid using these devices.

DETAILED DESCRIPTION:
The use of herbal treatment, also called phytotherapies, or dietary supplements or specific food (herbs, food or dietary supplements HFDS) is very common and have been evaluated between 30 and 70%, depending on the population and the studies.However, few studies have been made to evaluate the risk of interaction with oncology treatment in real life. Some interaction are very well known by both patients and clinicians, like the inhibition of the cytochrome 3A4 by grapefruit or the induction of the CYP3A4 by Saint John's Wort. However, many other interactions have been demonstrated, like the inhibition of the CYP3A4 by goldenseal extracts (among many others) although this is frequently used phytotherapy, both over the counter or "prescribed" by herb specialists.

This study aims at demonstrating that a smartphone or tablet application could be used to prevent significant interaction between phytotherapy or food or dietary supplements with anticancer treatments.

The application is used to collect data prospectively that will be analysed for interaction retrospectively. The interactions between phytotherapy have been classified in 4 categories :

* likely (clinically relevant data in the literature between the herb and the anticancer treatment either directly or through documented CYP interaction)
* possible (animal model or in vitro data in favor of an interaction)
* unlikely (clinical data or animal model or in vitro data in favor of no interaction)
* unknown (no data available or data from that could not allow a conclusion due to its poor quality or an ambiguous conclusion) The investigators aim at measuring the proportion of "likely" herb-drug interaction (or dietary supplement or food) in a population of patients followed and treated for a cancer, either local or metastatic.

The investigators also aim at characterizing the population, quantifying the proportion of patients taking HFDS and, to measure the proportion of "possible" herb-drug interaction.

ELIGIBILITY:
Inclusion Criteria:

* Men or women over 18 years old
* Subject currently receiving a treatment for cancer or who has a planned treatment (radiotherapy, surgery, chemotherapy, hormonotherapy, targeted therapy or other procedure)

Exclusion Criteria:

* The subject is not able to read
* The subject is not using any herb, food or dietary supplement with a daily consumption.
* The subject refuses to be part of the study
* The subject does not know the name of the anticancer therapy that he receives.
* The subject does not know if he uses either phytotherapy, specific food consumed daily or dietary supplements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of patient is composed of patient treated for different kind of cancer and which are using daily HFDS
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-13 (Actual); Primary Completion 2019-11-10 (Estimated); Study Completion 2019-11-11 (Estimated)

PRIMARY OUTCOMES:
Rate of interaction between HFDS (herb food and dietary supplements) and anticancer drugs whith a level of evidence graded as "likely" (clinical evidence) in a cohort of cancer patient using at least 1 HFDS daily. | 1 day
  Measure of the rate of patients having a consumption of at least 1 phytotherapy, aspecific food (which is a specific ingredient that is eaten daily, like daily consumption of grapefruit juice or green tea) or a dietary supplement and having a likely interaction (justified through a clinically proven cytochrome interaction or direct interaction) with their anticancer treatment. The interaction could be through an inhibition of a major CYP in the metabolism of the chemotherapy. Each potential interaction will be searched in the literature.
  Anticancer treatments include chemotherapy, targeted therapies, hormonotherapies, radiotherapy or surgery.

SECONDARY OUTCOMES:
Rate of patients using HFDS | 1 day
Description of the population using HFDS (age, primory tumor, tumor stage : local or metastasis, | 1 day
Rate of interaction between HFDS and anticancer drugs whith a level of evidence graded as "possible" (clinical evidence) in a cohort of cancer patient using at least 1 HFDS daily. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Mir, MD-PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Centre d'Investigation Clinique Paris-Est, Paris, France